CLINICAL TRIAL: NCT07099586
Title: Assessment of Serum Concentrations of Vitamin B12, Folic Acid, and Vitamin D in Women of Reproductive Age to Determine Recommended Supplementation Doses in the Preconception Period and During Pregnancy
Brief Title: Vitamin B12, Folic Acid, and Vitamin D Status in Women of Reproductive Age
Status: Recruiting | Type: Observational
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Nikolina Penava, Principal Investigator, University of Mostar
Other Study IDs: SUM-VITB12-FOL-D-2024
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Vitamin d, Vitamin B 12 and Folic Acid Concentrations; Micronutrient Status in Women of Reproductive Age; Vitamin Status Assessment
Keywords: vitamin B12; vitamin D; folic acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of Reproductive Age: This cohort includes women aged 18 to 49 years who are undergoing blood sampling for analysis of serum concentrations of vitamin B12, folic acid, and vitamin D. No interventions are administered. This is an observational, cross-sectional study.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — This is an observational study. No intervention will be administered. Participants will provide blood samples for micronutrient analysis.

SUMMARY:
This cross-sectional observational study aims to assess serum concentrations of vitamin B12, folic acid, and vitamin D in women of reproductive age in Herzegovina. The study is led by Professor Vajdana Tomić, MD, PhD, who serves as the Principal Investigator, at the Faculty of Health Studies, University of Mostar, Bosnia and Herzegovina. The goal is to determine whether current international supplementation guidelines reflect the actual micronutrient status of this population. A total of 360 women aged 18-49 will be enrolled between December 2024 and December 2025 after providing informed consent. The findings will inform population-specific recommendations for micronutrient supplementation during the preconception period and pregnancy.

The study will be conducted at the Faculty of Health Studies, University of Mostar, Bosnia and Herzegovina.

DETAILED DESCRIPTION:
Micronutrient intake-particularly vitamin B12, folic acid, and vitamin D-is essential during the preconception period and pregnancy to support fetal growth and reduce the risk of adverse outcomes such as preterm birth, low birth weight, and congenital anomalies. However, excessive intake may carry potential risks, including epigenetic changes, insulin resistance, and increased incidence of childhood asthma and obesity. Additionally, folic acid may mask underlying vitamin B12 deficiency, delaying diagnosis and increasing the risk of neurological complications.

This cross-sectional study addresses the lack of region-specific data on micronutrient status among women of reproductive age in Herzegovina. Although international guidelines provide general recommendations, they may not reflect the actual needs of this population. The study aims to evaluate the prevalence of micronutrient deficiency, adequacy, or excess to guide the development of evidence-based, locally adapted supplementation strategies.

A total of 360 women aged 18 to 49 will be enrolled between December 1, 2024, and December 1, 2025, after providing informed consent. Blood samples will be collected and centrifuged, and serum concentrations of vitamin B12, folic acid, and vitamin D will be measured using chemiluminescent microparticle immunoassays (CMIA) on the Alinity ci platform (Abbott Diagnostics). The study will be conducted in three phases: (1) participant recruitment and sample collection, (2) laboratory analysis and statistical evaluation using MedCalc software, and (3) preparation and publication of results in a peer-reviewed journal. The findings are expected to support more personalised and rational approaches to micronutrient supplementation in women planning pregnancy or who are already pregnant.

.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18-49 years)
* Informed consent obtained

Exclusion Criteria:

* diabetes (Type I or II)
* epilepsy
* oncological diseases, inflammatory bowel disease
* supplementation with vitamin B12, folic acid, or vitamin D within the last 3 months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes approximately 360 women aged 18 to 49 years from the Herzegovina region who participate after providing written informed consent. All participants are being screened according to defined inclusion and exclusion criteria. The study focuses on assessing serum concentrations of vitamin B12, folic acid, and vitamin D to support the development of population-specific supplementation guidelines for the preconception period and pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of vitamin B12 | At enrollment (single visit)
  Measured in serum samples using Alinity i immunoassay system.
Serum concentration of folic acid | At enrollment (single visit)
  Measured in serum samples using Alinity i immunoassay system.
Serum concentration of vitamin D | At enrollment (single visit)
  Measured in serum samples using Alinity i immunoassay system.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mostar, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and institutional policy limitations. All data will be analyzed and presented in aggregate form only, without identifying individual participants.